CLINICAL TRIAL: NCT01111162
Title: Evaluating the Safety and Immunogenicity of an Inactivated Swine-Origin H1N1 Influenza Vaccine in HIV-1 Infected Patients
Brief Title: H1N1 Influenza Vaccine Immunogenicity in HIV-1 Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Pablo Tebas, Professor of Medicine, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Upenn HIV-H1N1-001
Record Dates: First submitted 2010-04-13; First posted 2010-04-27 (Estimated); Results first posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: HIV Infections
Keywords: HIV; H1N1 vaccination; HIV infected individuals
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine (Experimental): Novartis unadjuvanted inactivated S-OIV H1N1 influenza vaccine 15 mcg administered as single-0.5mL (15mcg) injection intramuscularly into one of the subject's deltoid muscles
  Interventions: Biological: H1N1 vaccination

INTERVENTIONS:
Biological: H1N1 vaccination — Novartis unadjuvanted inactivated S-OIV H1N1 influenza vaccine 15 mcg administered as single-0.5mL (15mcg) injection intramuscularly into one of the subject's deltoid muscles

SUMMARY:
The overall goal of this study is to study influenza vaccine responses in HIV infected individuals. Immunocompromised individuals require special protection from influenza, but may not respond appropriately to the standard killed vaccine. Patients who receive the H1N1 flu vaccine as part of their standard of care will be asked to donate blood samples for immunologic studies. These studies will determine whether participants were able to produce the appropriate antibodies to the vaccine and possibly identify predictors of vaccine responsiveness.

Our hypothesis is that vaccine responsiveness to the new H1N1 influenza vaccine will be compromised in HIV infected patients.

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed diagnosis of HIV-1 infection as documented by any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry or any measurable HIV RNA viral load in the chart. Serum HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
2. > 18 years
3. Able to understand and comply with planned study procedures.
4. Provides written informed consent prior to initiation of any study procedures.
5. Subject should be 1) on stable antiretroviral therapy as outlined in the DHHS treatment guidelines for HIV-1 infected individuals OR 2) not on antiretroviral therapy and not intending to start treatment within the next 30 days.

Exclusion Criteria:

1. Has a known allergy to eggs or other components in the vaccines (these may include, but are not limited to: gelatin, formaldehyde, octoxinol and chicken protein).
2. Has a history, in the opinion of the site investigator, of severe reactions following previous immunization with seasonal TIV.
3. Participation in a novel H1N1 influenza vaccine study in the past two years.
4. Proven history, by RT-PCR, of novel influenza H1N1 infection, or, has a positive influenza diagnostic testing since June 2009 (specificity to H1N1 not required) prior to study entry.
5. Received any other live licensed vaccine within 4 weeks or inactivated licensed vaccine within 1 week prior to study entry.
6. Scheduled administration of any live virus vaccine or inactivated vaccine at or between entry and the Day 21 visit. NOTE: Live or inactivated vaccines expected to be administered between study entry and the Day 21 visit should be excluded to prevent potential interference with immunogenicity responses and confounding safety results. Regular seasonal flu vaccination will be allowed if is separated more than 7 days from the administration of the H1N1 vaccine.
7. Received a non-licensed agent (vaccine, drug, biologic, device, blood product, or medication) within 4 weeks prior to vaccination in this study
8. An acute illness and/or an oral temperature greater than or equal to 100.0 degrees F within 24 hours prior to study entry.
9. Use of anti-cancer chemotherapy or radiation therapy within the preceding 36 months of study enrollment, or has immunosuppression as a result of an underlying illness or treatment (other than HIV-1 infection).
10. Active neoplastic disease (excluding non-melanoma skin cancer, and HPV-related cervical dysplasia, CIN grades 1, 2 or 3).
11. Long term use of glucocorticoids, including oral or parenteral prednisone or equivalent (more than 2.0 mg/kg per day or more than 20 mg total dose) for more than 2 consecutive weeks (or 2 weeks total) in the past 3 months, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the past 3 months (nasal and topical steroids are allowed).
12. Received immunoglobulin or other blood products
13. Current diagnosis of uncontrolled major psychiatric disorder.
14. History of Guillain-Barré Syndrome in the subject or subject's family (parents, siblings, half siblings, or children).
15. Any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-12; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Tebas, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania. Clinical Trials Unit, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Tebas P, Frank I, Lewis M, Quinn J, Zifchak L, Thomas A, Kenney T, Kappes R, Wagner W, Maffei K, Sullivan K; Center for AIDS Research and Clinical Trials Unit of the University of Pennsylvania. Poor immunogenicity of the H1N1 2009 vaccine in well controlled HIV-infected individuals. AIDS. 2010 Sep 10;24(14):2187-92. doi: 10.1097/QAD.0b013e32833c6d5c. PMID 20616698

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at the MacGregor Clinic of the Hospital of the University of Pennsylvania in Philadelphia, Pennsylvania, USA, between the months of November and January 2009-2010. All patients signed an informed consent. The study was approved by the University of Pennsylvania institutional review board .
Groups:
- Vaccine Arm (Single Arm): 15 µg dose of the monovalent, unadjuvanted, inactivated, split virus H1N1 vaccine (Novartis, Basel, Switzerland).
Period: Overall Study
Arm/Group | Vaccine Arm (Single Arm)
Started | 120
Completed | 120
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Vaccination Group (Single Arm Study): All participants
Arm/Group | Vaccination Group (Single Arm Study)
Number analyzed (Participants) | 120
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [40 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 113
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 81
  White | 37
  More than one race | 0
  Unknown or Not Reported | 0
Percentage of Participants at Baseline with HAI assay titers ≥ 1:40 [Number; unit: percentage of participants] | 25

OUTCOME MEASURES:

1. Primary Outcome: Safety
Description: To assess the safety of inactivated swine-origin H1N1 influenza vaccine in HIV-1 infected individuals (received as part of standard of care).
  Safety was assessed via
  1. Adverse Events of Grade 3 or higher of abnormal laboratory values, signs and symptoms or diagnoses.
  2. Solicited local AEs, including pain, tenderness, redness, and swelling post each vaccination. Solicited systemic AEs, including feverishness, malaise, body aches (exclusive of the injection site), nausea, and headache post each vaccination.
Time Frame: 21-28 days
Measure: Number; unit: percentage of participants
Arm/Group | Vacinees
Number analyzed (Participants) | 120
percentage of participants
  Pain | 22
  Redness | 3
  Induration | 0
  Tenderness | 18
  Ecymosis | 0
  Headache | 16
  Malaise | 19
  Myalgia | 18
  Nausea | 4
  Chills | 3
  Vomiting | 1
  Fever | 1

2. Primary Outcome: Immunogenicity
Description: Immunologic response, defined as HAI titer ≥ 1:40, at 21 days after vaccine dose.
Time Frame: 21-28 days
Population: Among the 90 participants without evidence of previous exposure to H1N1, only 61% [95% confidence interval (CI) 51-71] developed protective titers by week 3 of the study (seroconversion rate).
Measure: Number (95% Confidence Interval); unit: percentage of seroconversion
Arm/Group | Vaccine Arm (Single Arm)
Number analyzed (Participants) | 90
percentage of seroconversion | 61 [51 to 71]

ADVERSE EVENTS:
Time Frame: Duration of the study (21-28 days)
Description: Serious adverse events include all Grade 3 or greater adverse events
Arm/Group | Vaccine Arm (Single Arm)
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 31/120
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine Arm (Single Arm) (N=120)
Pain at Injection Site (General disorders) | 26 — Administration site reaction
Redness at Injection Site (General disorders) | 4 — Administration site reaction
Tenderness at Injection Site (General disorders) | 22 — Administration site reaction
Headache (General disorders) | 19 — Systemic site reaction
Malaise (General disorders) | 23 — Systemic site reaction
Myalgia (General disorders) | 22 — Systemic site reaction
Nausea (General disorders) | 5 — Systemic site reaction
Chills (General disorders) | 3 — Systemic site reaction
Vomiting (General disorders) | 1 — Systemic site reaction
Fever (General disorders) | 1 — Systemic site reaction

LIMITATIONS AND CAVEATS:
Single Arm Study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No